CLINICAL TRIAL: NCT07278687
Title: LATA-IBD Trial a Laparoscopic and Transanal IPAA-surgery Trial.
Brief Title: LATA-IBD TRIAL a Controlled Feasibility Study for the Introduction of Transanal Minimally Invasive IPAA-Surgery. Evaluation of Operative Results and Bowel Function After Introducing Transanal IPAA-surgery to Replace Conventional Laparoscopic IPAA-surgery.
Acronym: LATA-IBD
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Bjarne Melvas, Senior consultant,, Sahlgrenska University Hospital
Other Study IDs: Dnr 2024-03692-02
Record Dates: First submitted 2025-11-22; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis (Disorder); Familial Adenomatous Polyposis (FAP)
Keywords: ulcerative colitis; laparoscopy; transanal surgery; pelvic pouch
MeSH Terms: conditions — Colitis, Ulcerative; Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 22 Patients operated with transanal laparoscopic IPAA: Proaspecticely collected data with paper case report form
- 17 Patients operated with conventional laparoscopic IPAA: Retrospectively collected data from medical records

SUMMARY:
This study compares the operative and functional outcomes of adding a transanal pathway to laparoscopic pelvic pouch surgery. The transanal pathway enables the surgeon to have better control when dividing the rectum and it may improve visualization in pelvic dissection. This could decrease the need for conversion to open surgery, reduce complications, postoperative pain, hospital stay and improve bowel function after surgery. The study compares two consecutive groups of patients at a single institution. The transanally operated group consists of 22 patients with prospectively collected data between 2018-2020 and the traditional laparoscopic group consists of 17 patients with retrospectively collected data operated between 2015-2016. Inclusion criteria for the transanal group were patients over 18 years with either ulcerative colitis or familial adenomatous polyposis who were possible to operate with laparoscopic surgery and who had signed an informed consent.

The studys primary objective is to investigate if there is a difference in the frequency of conversions to open surgery or anastomotic leakage of the anastomosis between the pelvic pouch and the anal canal. Secondary objectives are mortality, bleeding, operative time, complications, reoperations, hospital stay, readmissions to hospital and bowel function two years after surgery.

DETAILED DESCRIPTION:
Study Design This is a prospective feasibility study comparing consecutive patients undergoing ta-IPAA with a historical cohort of patients treated with lap-IPAA at the same institution.

Endpoints The primary endpoints were conversion rate and anastomotic leakage rate. Conversion was defined as the need for laparotomy before pouch construction and/or specimen extraction, or the requirement to extend or alter the initial incision during pouch construction. Anastomotic leakage was defined and graded according to the International Study Group of Rectal Cancer (18).

Secondary endpoints included mortality, intraoperative bleeding, operative time, postoperative complications (graded according to the Clavien Dindo classification (19)), reoperations, readmissions, length of hospital stay and pouch function. Pouch function was assessed using the Öresland score (OS) (20) two years after surgery. The OS consists of 11 parameters measuring bowel function after IPAA and ranges from 0-15 (higher scores indicate worse function). Scores ≥8 are associated with impaired pouch function and reduced quality of life. Pouch failure was defined as the need for a diverting stoma or excision of the pouch.

Data collection Study data were collected prospectively using a paper case report form (CRFs) completed at predefined time points: preoperatively, intraoperatively, at hospital discharge and 3, 6, 12 and 24 months after ta-IPAA. For the historical control group, data were retrieved retrospectively from medical records. Intraoperative data were excluded from the lap-IPAA group, as these could not be reliably retrieved.

Training The surgical team consisted of three colorectal surgeons and experienced operating room nurses, all with prior expertise in laparoscopic Total Mesorectal Excision (TME) and IPAA-surgery. The team underwent formal training in taTME-surgery, including participation in dedicated courses, observational visits and on-site proctoring by an international center with significant experience in ta-IPAA.

Surgical Procedure The procedure began with takedown of the loop ileostomy. If mesenteric length was sufficient, the pouch was constructed immediately; otherwise, pouch construction was delayed until the abdominal phase, using either a midline or suprapubic incision. The abdomen was insufflated, and the mesentary was freed from adhesions and the duodenum. Mesenteric lengthening techniques were applied as required before constructing the ileal pouch.

Rectal dissection was performed in a modified TME plane, remaining closer to the rectum, particularly anteriorly, for the first two-thirds of the dissection. The transanal approach was used for the final third, employing standard equipment including the GelPOINT Path Transanal Access Platform®, Lone Star retractor®, and AirSeal® System. Dissection was performed with monopolar cautery, and the purse-string suture was placed with 3-0 V-Loc®. The rectum was extracted transanally or, if necessary, via an abdominal incision. The ileoanal anastomosis was constructed with a circular stapler, and a diverting stoma was created at the previous ileostomy site. (21)

ELIGIBILITY:
Inclusion Criteria

* 18 years and over.
* UC or FAP.
* Fit for laparoscopic IPAA-surgery
* Signed informed consent.

Exclusion Criteria

- Not meeeting inclusion criteria above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients aged >18 years with a diagnosis of ulcerative colitis (UC) or familial adenomatous polyposis (FAP) scheduled for lap-IPAA between 2018 and 2020 at Sahlgrenska University Hospital were invited to participate. A minimum sample size of 20 patients was considered sufficient to evaluate the feasibility of introducing the ta-IPAA technique. For comparison, a historical control group of 17 patients who underwent lap-IPAA between 2015 and 2016 was identified.
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Conversion rate to open surgery | During surgery
  Rate of patients with abdominal incision before pouch construction or changed or extended abdominal incision during pouch construction.
Anastomotic leakage rate | Within 24 months after surgery
  Rate of anastomotic leakage as defined by the international study group of cancer. A defect of the intestinal wall at the anastomotic site (including suture and staple lines of neorectal reservoirs) leading to a communication between the intra- and extraluminal compartments.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna de la Croix, Associate professor, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital/East department, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data may be shared if needed but only if the secrecy of the patients is maintained. Data will be presented as group data in the publication.

REFERENCES:
- [Background] Deng SX, Brar MS, Yang ML, Park JJ, de Buck van Overstraeten A. Functional outcomes of transanal ileal pouch anal anastomosis in patients with ulcerative colitis: inverse-probability weighing analysis of a single-center cohort. J Gastrointest Surg. 2025 Oct;29(10):102189. doi: 10.1016/j.gassur.2025.102189. Epub 2025 Aug 13. PMID 40816645
- [Background] Stephens IJB, Byrnes KG, Burke JP. Transanal ileal pouch-anal anastomosis: A systematic review and meta-analysis of technical approaches and clinical outcomes. Langenbecks Arch Surg. 2024 May 6;409(1):153. doi: 10.1007/s00423-024-03343-7. PMID 38705912
- [Background] de Buck van Overstraeten A, Mark-Christensen A, Wasmann KA, Bastiaenen VP, Buskens CJ, Wolthuis AM, Vanbrabant K, D'hoore A, Bemelman WA, Tottrup A, Tanis PJ. Transanal Versus Transabdominal Minimally Invasive (Completion) Proctectomy With Ileal Pouch-anal Anastomosis in Ulcerative Colitis: A Comparative Study. Ann Surg. 2017 Nov;266(5):878-883. doi: 10.1097/SLA.0000000000002395. PMID 28742696
- [Background] Violante T, Broccard SP, Novelli M, Stocchi L, Colibaseanu DT, DeLeon MF, Behm KT, Mishra N, Larson DW, Merchea A. Comparative analysis of robotic, laparoscopic, and open ileal pouch-anal anastomosis outcomes: retrospective cohort study. BJS Open. 2025 Jul 1;9(4):zraf084. doi: 10.1093/bjsopen/zraf084. PMID 40742352